CLINICAL TRIAL: NCT00880308
Title: A Phase I, Multicenter, Open-label, Dose-escalation Study of Oral LDE225 in Patients With Advanced Solid Tumors
Brief Title: Dose Finding and Safety of Oral LDE225 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLDE225X2101; 2008-005603-26 (EudraCT Number)
Record Dates: First submitted 2009-04-09; First posted 2009-04-13 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2014-12

CONDITIONS: Advanced Solid Tumor Cancers; Medulloblastoma; Basal Cell Carcinoma
Keywords: Advanced tumors; hedgehog; smoothened inhibitor
MeSH Terms: conditions — Medulloblastoma; Carcinoma, Basal Cell | interventions — sonidegib

ARMS (1):
- LDE225 (Experimental)
  Interventions: Drug: LDE225

INTERVENTIONS:
Drug: LDE225

SUMMARY:
This first-in-human dose-escalation study is to characterize the safety, tolerability, pharmacokinetics and pharmacodynamics of LDE225 given orally on a daily dosing schedule in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of advanced solid tumor (including •medulloblastoma and basal cell carcinoma)
* blood work criteria

Exclusion Criteria:

* patients with history of brain tumor (except recurrent medulloblastoma) or brain metastases
* positive HIV, hepatitis B or C
* impaired intestinal function
* impaired heart function
* pregnant or breast-feeding women

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2009-03; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
determine maximum tolerated dose of single agent LDE225 | 28 day cycles

SECONDARY OUTCOMES:
characterize safety and tolerability | 28 day cycles
characterize pharmacokinetics (PK) of single and repeated doses of LDE225 | 28 day cycles
assess preliminary anti-tumor activity | every other 28-day cycle

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (5):
- United States (2):
  - University of Pittsburgh Medical Center SC, Pittsburgh, Pennsylvania
  - Cancer Therapy & Research Center / UT Health Science Center InstituteForDrugDevelopment(5), San Antonio, Texas
- Novartis Investigative Site, Barcelona, Catalonia, Spain
- Novartis Investigative Site, Zurich, Switzerland
- Novartis Investigative Site, Leicester, United Kingdom

REFERENCES:
- See also: Results for CLDE225X2101 on Novartis Clinical Trials Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=12203